CLINICAL TRIAL: NCT04998006
Title: Exploring the Effects of Cannabinoids on Alcohol Consumption and the Microbiota-Gut-Brain Axis
Brief Title: Alcohol and Cannabis Co-Use and the Gut-Brain Axis
Acronym: FRACTAL
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Hollis Karoly, Associate Professor, University of Colorado, Denver
Other Study IDs: 24-2424; K23AA028238 (NIH)
Record Dates: First submitted 2021-06-30; First posted 2021-08-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-01

CONDITIONS: Cannabis Use; Alcohol Use; Inflammation
Keywords: Alcohol; Cannabis; Microbiome; Marijuana
MeSH Terms: conditions — Alcohol Drinking; Inflammation; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen description: whole blood will be collected, plasma will be retained, fecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall Study Cohort: Over a period of four weeks, participants completed two Phases (A and B) followed by two visits in our mobile laboratory (Visits A and B). The order of which was counterbalanced across participants so that approximately half of the participants completed Phase A/Visit A first, and the other half completed Phase B/Visit B first.
  Phase A involved 2 weeks of no cannabis use followed by a mobile laboratory session (Visit A), involving biological sample collection, neurobehavioral testing, and an alcohol self-administration task. Phase B involved 2 weeks of ad-libitum use of participant-preferred cannabis products, followed by a session in the mobile laboratory (Visit B) in which participants completed the same neurobehavioral tasks, biological sample collection, and alcohol self-administration task immediately following acute ingestion of preferred cannabis strain in participant homes.

SUMMARY:
This observational study aims to improve our understanding of how legal market cannabis use impacts acute and long-term alcohol use, the microbiota-gut-brain-axis (MGBA), and neurobehavioral alcohol use phenotypes such as impulsivity, impaired cognitive functioning, and craving, among individuals who regularly use both alcohol and cannabis. Over a period of one month, subjects will participate in this three-visit study. Blood samples will be collected to allow for the assessment of inflammatory markers and cannabinoids, a fecal sample will be collected to allow for the analysis of the gut microbiome, and participants will complete cognitive and impulsivity tasks and provide craving ratings during the course of an alcohol self-administration procedure. Subjects will also participate in two 14-day daily diary data collection periods between lab sessions. Daily diary data collection will be used to assess the effects of cannabis use on alcohol use and craving longitudinally.

DETAILED DESCRIPTION:
At present, the consumption of alcohol and alcohol use disorder (AUD) constitute a public health crisis. Due to the neurobiological complexity of AUD, the development of new treatments requires a deeper understanding of the molecular mechanisms underlying etiology and course of AUD. This includes the degree to which cannabis use may reduce or enhance harms of alcohol consumption through cannabinoid influence on gut and immune functions. One potential mechanism through which cannabinoids may exert beneficial effects in heavy drinkers is through their role in modulating the gut microbiome and immune system, which have been found to be disrupted by alcohol. However, it is also possible that cannabinoids, specifically delta-9-Tetrahydrocannabinol (THC), may confer harms in heavy drinkers by enhancing the intoxicating effects of alcohol. The current study will be the first to explore the acute and long-term effects of cannabis on alcohol use and neurobehavioral phenotypes, including alcohol craving, impulsivity, and impaired cognition, as well as the impact of cannabinoids on the microbiota-gut-brain-axis (MGBA) in human non-treatment-seeking, regular-cannabis-using heavy drinkers.

This study examines the effects of legal market cannabis on acute and long-term alcohol use, (specifically the effects of alcohol and cannabis use on gut microbiome and inflammatory markers in the blood) in a 4-week, observational design using both traditional and mobile lab settings, as well as self-report, daily diary methodology. Participants will complete two Phases (A and B) following by two visits to our mobile laboratory (Visits A and B), the order of which will be counterbalanced across participants so that half of participants will complete phase A/visit A first, and the other half will complete Phase B/Visit B first. Phase A involves 2 weeks of no cannabis use followed by a mobile lab session (Visit A), involving biological sample collection, neurobehavioral testing and an alcohol self-administration task. Phase B involves 2 weeks of ad lib use of participant preferred cannabis product, followed by a session in the mobile lab session (Visit B) in which participants will complete the same neurobehavioral tasks, biological sample collection, and alcohol self-administration task immediately following acute ingestion of preferred cannabis strain in participant homes.

ELIGIBILITY:
Inclusion Criteria:

1. 21-60 years of age
2. Able to provide consent
3. Heavy drinker, defined as: for men, consuming more than 4 drinks on any day or more than 14 drinks per week OR, for women, consuming more than 3 drinks on any day or more than 7 drinks per week over the last 3 months.
4. Regular legal-market cannabis smoker, defined as using smoked flower cannabis obtained from a dispensary at least 3 days per/week over the past 3 months
5. Willing to abstain from cannabis use for 14 days
6. We are prioritizing the recruitment of participants in the Fort Collins/Loveland area

Exclusion Criteria:

1. Daily tobacco use*** (Vape and Hooka included)
2. Actively seeking treatment for alcohol use disorder or other substance use disorder
3. Females cannot be pregnant, breastfeeding or trying to become pregnant
4. Meet criteria for psychotic, bipolar or major depressive disorder with suicidal ideation, or history of these disorders
5. Immune-relevant disease (e.g., osteoarthritis, HIV, cancer, recent infection, other autoimmune disorder) or currently taking an immune-modulating medication***
6. Current use of psychotropic medications (except anti-depressants )
7. Report illicit drug use in past 60-days or fail drug screen
8. Major medical condition that contraindicates the consumption of alcohol or cannabis.
9. Use of an antibiotic medication in the past 3 months
10. Current GI disorder including: inflammatory bowel disease, irritable bowel disease, diverticular disease, peptic ulcer/gastritis and gastroesophageal reflux disease.
11. Use of probiotic or supplement drinks at least once per week over the last 3 months

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Acute alcohol consumption | Change over two time points: Session A (alcohol administration only) and Session B (alcohol administration + ad-libitum cannabis administration). Sessions A and B are 2 weeks apart.
  Total number of drinks consumed (out of 4) in a one-hour period.
Impulsivity Cognition: Stop Signal Task | Change over two time points (Session A [alcohol administration only] and Session B [alcohol administration + ad-libitum cannabis administration]) 2 weeks apart: Pre-alcohol/cannabis consumption, Post-alcohol/cannabis consumption
  This task requires responding quickly to "go" signals, and occasionally inhibiting those responses when a "stop" signal is displayed.
Daily alcohol consumption | Change over two consecutive 14-day daily time periods
  Two 14-day daily data collection periods using self-report of alcohol craving and amount of alcohol consumed
Inflammation | Change over two time points (Session A [alcohol administration only] and Session B [alcohol administration + ad-libitum cannabis administration]) 2 weeks apart
  Test levels of inflammation (panel of inflammatory cytokines) at Session A (following 2 weeks of no cannabis use) and Session B (following 2 weeks of ad lib cannabis use).
Gut microbiota | Change over two time points (Session A [alcohol administration only] and Session B [alcohol administration + ad-libitum cannabis administration]) 2 weeks apart.
  Outcomes of interest include gut bacterial diversity and composition. Gut microbiome data from Session A will be compared with gut microbiome data from Session B.

SECONDARY OUTCOMES:
Change in Alcohol Craving (Visual-Analog Scale | Change over two time points: Session A (alcohol administration only) and Session B (alcohol administration + ad-libitum cannabis administration). Sessions A and B are 2 weeks apart
  Test differences in alcohol craving using Visual Analog Scale in laboratory sessions in which only alcohol is consumed (Session A) and in which cannabis is self-administered prior to alcohol administration (Session B). Possible values range from 0-10, with higher scores indicating greater alcohol craving.
NIH Toolbox Flanker Test | Change over two time points (Session A [alcohol administration only] and Session B [alcohol administration + ad-libitum cannabis administration]) 2 weeks apart: Pre-alcohol/cannabis consumption, Post-alcohol/cannabis consumption
  This task requires participants to sustain attention on a stimulus while inhibiting attention to stimuli flanking it.
Intestinal permeability | Change over two time points (Session A [alcohol administration only] and Session B [alcohol administration + ad-libitum cannabis administration]) 2 weeks apart
  Test levels of recent intestinal permeability measured in blood at Session A (following 2 weeks of no cannabis use) and Session B (following 2 weeks of ad lib cannabis use).
The Alcohol Purchase Task (APT) | Change between reward value of alcohol when cannabis is on board (session B) compared to when it is not (session A). This task will also be administered at baseline (when not intoxicated) to compare sober state-level alcohol reward
  The APT is a is a well-validated, easy-to-administer measure that will be given at baseline and multiple times during session A and B. This task measures the reinforcing value of alcohol using simulated marketplace survey techniques (i.e. - how many drinks would you purchase if they cost 50 cents?)

OTHER OUTCOMES:
Exploratory: Daily Follow-up Messages | Brief self-report from participants on cannabis use, exercise, and mood in the past 24 hours.
  Change over two consecutive 14-day daily time periods.
Plasma Gamma-Glutamyl Transferase (GGT) | Change over two time points (Session A [alcohol administration only] and Session B [alcohol administration + ad-libitum cannabis administration]) 2 weeks apart
  Test levels of recent liver inflammation (GGT) at Session A (following 2 weeks of no cannabis use) and Session B (following 2 weeks of ad lib cannabis use). (Not collected)
Change in Rey Auditory Verbal Learning Test (RAVLT) | Change over two time points (Session A [alcohol administration only] and Session B [alcohol administration + ad-libitum cannabis administration]) 2 weeks apart: Pre-alcohol/cannabis consumption, Post-alcohol/cannabis consumption
  The RAVLT is a neuropsychological assessment designed to evaluate verbal memory in adult patients. The RAVLT can be used to evaluate the nature and severity of memory dysfunction and to track changes in memory function over time.

CONTACTS AND LOCATIONS:
Overall Officials: Hollis C. Karoly, PhD, Principal Investigator — CU Anschutz School of Medicine
Locations (1):
- CU Anschutz School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will submit all de-identified individual level phenotypic human subjects data from this project to the NIAAA data archive. The project also involves collection of human specimens (fecal samples) which will generate non-human genomic data. Specifically, the investigators plan to generate 122 (61 subjects x 2 timepoints) human gut microbiota metagenomes (i.e., gut microbiome). Deidentified genomic data from microbiome assays (and relevant phenotypic data) will be submitted to the database of Genotypes and Phenotypes (dbGaP).
Time Frame: Human phenotypic data will be uploaded at least twice a year. Non-human genomes from fecal samples will be shared within 3 months of processing and genotyping all meta-genomes
Access Criteria: Data access through the National Institute of Mental Health Data Archive (NIAAA) and dbGaP.

REFERENCES:
- [Derived] Gowin JL, Stallsmith V, Weldon K, Dooley G, Karoly HC. Effects of legal-market cannabis and alcohol on verbal learning and memory. Psychopharmacology (Berl). 2025 Sep 25. doi: 10.1007/s00213-025-06882-z. Online ahead of print. PMID 40996525